CLINICAL TRIAL: NCT06830005
Title: Validating Osteoporosis Detection in Rho AI Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-1832; A536100 (Other: UW Madison); Protocol Version (Other: UW Madison)
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Osteopenia or Osteoporosis
Keywords: orthopedic surgery; screening
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Experimental Detection of Osteoporosis (Experimental)
  Interventions: Device: Rho AI software

INTERVENTIONS:
Device: Rho AI software — Rho is a AI enabled opportunistic pre-screening computer-aided detection and notification software for low bone mineral density.

SUMMARY:
To assess the effectiveness of 16bit's Rho AI (artificial intelligence) software at identifying known cases of osteoporosis. 800 de-identified images from January 2007 to January 2024 will be accessed to test the software prospectively.

DETAILED DESCRIPTION:
Osteoporosis is underrecognized and undertreated in the orthopedic surgery patient population. Osteoporosis is diagnosed by dual-energy x-ray absorptiometry which is costly and imparts radiation. Preoperative radiographs are universally obtained in orthopedic surgery patients, however up to this point radiographs have not been able to diagnose osteoporosis. This software program is a new technology that is able to leverage radiographs to opportunistically screen for osteoporosis.

The study team will identify applicable patient records from medical record review, and Radius will de-identify the x-ray images. The de-identified images will be run through the Rho AI program to identify osteoporosis or osteopenia, and a report will be generated to summarize the program's findings.

ELIGIBILITY:
Inclusion Criteria:

* images from people who have undergone total joint arthroplasty
* images from people who have undergone spine fusion

Exclusion Criteria:

-

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
AI Predicted Osteoporosis Score | through study completion (data collected up to 1 month)
  Osteoporosis score is a T-score where -1.0 and above: Normal bone density, -1.0 to -2.5: Osteopenia (low bone mass), -2.5 and below: Osteoporosis

CONTACTS AND LOCATIONS:
Overall Officials: James Bernatz, MD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- UW School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No